CLINICAL TRIAL: NCT01953978
Title: The Effect of Dexamethasone in Combination With Paracetamol and Ibuprofen as Adjuvant, Postoperative Pain After Herniated Disc Surgery
Brief Title: The Effect of Dexamethasone in Combination With Paracetamol and Ibuprofen on Postoperative Pain After Spine Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Rikke Vibeke Nielsen, MD, MD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM-RS-2012; 2012-004181-18 (EudraCT Number)
Record Dates: First submitted 2013-09-26; First posted 2013-10-01 (Estimated); Last update posted 2015-10-27 (Estimated); Status verified 2015-10

CONDITIONS: Pain
Keywords: Pain; Analgesia; Postoperative; Dexamethasone; Spine surgery
MeSH Terms: conditions — Pain; Agnosia | interventions — Dexamethasone; Morphine; Ondansetron; Acetaminophen; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dexamethasone (Active Comparator): * Intravenous administration of dexamethasone 16 mg (concentration 4 mg/ml, volume 4 ml) immediately after endotracheal intubation
  * Morphine. Patient controlled intravenous morphine (PCA-pump), bolus 2.5 mg, lock-out-time 10 minutes. Concentration : Morphin 1 mg/ml.
  * Zofran 4 mg iv in case of moderate to severe nausea, supplemented by Zofran 1 mg iv if needed
  * Tablet Paracetamol 1 g orally and tablet Ibuprofen 400 mg orally. Both 1 hour preoperatively and every 6 hours after extubation time during the first 48 hours.
  Interventions: Drug: Dexamethasone; Drug: Morphine; Drug: Zofran; Drug: Paracetamol; Drug: Ibuprofen
- Placebo (Placebo Comparator): * Intravenous administration of isotonic sodium chloride (concentration 9 mg/ml, volume 4 ml) immediately after endotracheal intubation
  * Morphine. Patient controlled intravenous morphine (PCA-pump), bolus 2.5 mg, lock-out-time 10 minutes. Concentration : Morphin 1 mg/ml.
  * Zofran 4 mg iv in case of moderate to severe nausea, supplemented by Zofran 1 mg iv if needed
  * Tablet Paracetamol 1 g orally and tablet Ibuprofen 400 mg orally. Both 1 hour preoperatively and every 6 hours after extubation time during the first 48 hours.
  Interventions: Other: Placebo; Drug: Morphine; Drug: Zofran; Drug: Paracetamol; Drug: Ibuprofen

INTERVENTIONS:
Drug: Dexamethasone — Intravenous administration of dexamethasone 16 mg (concentration 4 mg/ml, volume 4 ml) immediately after endotracheal intubation
  Arms: Dexamethasone
Other: Placebo — Intravenous administration of isotonic sodium chloride (concentration 9 mg/ml, volume 4 ml) immediately after endotracheal intubation
  Arms: Placebo
Drug: Morphine — Morphine. Patient controlled intravenous morphine (PCA-pump), bolus 2.5 mg, lock-out-time 10 minutes. Concentration : Morphin 1 mg/ml.
Drug: Zofran — Zofran 4 mg iv in case of moderate to severe nausea, supplemented by Zofran 1 mg iv if needed
Drug: Paracetamol — Tablet Paracetamol 1 g orally, 1 hour preoperatively and every 6 hours after extubation time during the first 48 hours.
Drug: Ibuprofen — Tablet Ibuprofen 400 mg orally, 1 hour preoperatively and every 6 hours after extubation time during the first 48 hours.

SUMMARY:
The analgesic effect of dexamethasone is not well described, but studies have shown that dexamethasone can be a safe part of a multimodal analgesic strategy after surgery. Our purpose is to investigate if dexamethasone in combination with paracetamol and ibuprofen has an increased analgesic effect compared to paracetamol and ibuprofen alone, on postoperative pain after spine surgery. Our hypothesis is that dexamethasone can reduce postoperative pain and reduce opioidconsumption and side effects compared to placebo.

DETAILED DESCRIPTION:
The analgesic effect of dexamethasone is not well described, but studies have shown that an intermediate dosis of dexamethasone (0.11-0.2 mg/kg) can be a safe part of a multimodal analgesic strategy after surgery. Dexamethasone has an opioid-sparing effect and reduces pain during rest and mobilisation. Our purpose is to investigate if dexamethasone in combination with paracetamol and ibuprofen has an increased analgesic effect compared to paracetamol and ibuprofen alone, on postoperative pain after herniated disk surgery. Our hypothesis is that dexamethasone can reduce postoperative pain and reduce opioidconsumption and side effects compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing lumbar disc surgery in general anaesthesia.
* Patients who have given their written consent to participate and understand the contents of the protocol.
* ASA 1-3.
* BMI > 18 og < 40.
* Fertile women need a negative HCG urine test.

Exclusion Criteria:

* Patients who cannot cooperate to the study.
* Patients who do not speak and/or understand Danish.
* Fertile women with a positive HCG urine test.
* Allergy to the drugs used in the trial.
* Alcohol or medicine abuse, assessed by investigator.
* Patients who have had spine surgery before.
* Daily use of strong opioids (morphine, ketobemidone, oxynorm, methadone, fentanyl)
* Daily oral steroid treatment.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2012-12; Primary Completion 2014-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Painscore during mobilization | 2-24 hours after extubation time.
  Painscore during active mobilization (VAS scale) defined by a standarized movement from recumbent position to sitting on the bedside at time 2, 4, 8, 12 and 24 hours, calculated as area under curve (AUC) from 2-24 hours after extubation time.

SECONDARY OUTCOMES:
Painscore during rest | 2-24 hours after extubation time
  Painscore during rest (VAS scale) at time 2, 4, 8, 12 and 24 hours, calculated as area under curve (AUC) from 2-24 hours after extubation time.
Morphine consumption | 0-24 hours after extubation time.
  Total morphine consumption 0-24 hours after extubation time, administered as patient controlled analgesia (PCA, bolus 2.5 mg, lockout 10 minutes).
Painscore during rest and mobilization | 48 hours after extubation time
  Painscore during rest and during active mobilization (VAS scale) at time 48 hours after extubation time.
Degree of nausea | 2, 4, 8, 12, 24 and 48 hours after extubation time
  Degree of nausea 2, 4, 8, 12, 24 and 48 hours after extubation time
Incidence of vomiting | 0-2, 2-4, 4-8, 8-12, 12-24 and 24-48 hours after extubation time.
  Total number of vomits 0-2, 2-4, 4-8, 8-12, 12-24 and 24-48 hours after extubation time.
Zofran consumption | 0-24 and 24-48 hours after extubation time.
  Consumption of Zofran (milligram) 0-24 and 24-48 hours after extubation time.
Degree of sedation | 2, 4, 8, 12, 24 and 48 hours after extubation time.
  Degree of sedation 2, 4, 8, 12, 24 and 48 hours after extubation time.
Quality of sleep | 24 hours after extubation time.
  Quality of sleep 24 hours after extubation time.

CONTACTS AND LOCATIONS:
Overall Officials: Rikke Soennichsen, MD, Principal Investigator — Glostrup University Hospital; Joergen B Dahl, MD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Glostrup University Hospital, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Nielsen RV, Fomsgaard J, Mathiesen O, Dahl JB. The effect of preoperative dexamethasone on pain 1 year after lumbar disc surgery: a follow-up study. BMC Anesthesiol. 2016 Nov 16;16(1):112. doi: 10.1186/s12871-016-0277-z. PMID 27852230
- [Derived] Nielsen RV, Siegel H, Fomsgaard JS, Andersen JDH, Martusevicius R, Mathiesen O, Dahl JB. Preoperative dexamethasone reduces acute but not sustained pain after lumbar disk surgery: a randomized, blinded, placebo-controlled trial. Pain. 2015 Dec;156(12):2538-2544. doi: 10.1097/j.pain.0000000000000326. PMID 26270586